CLINICAL TRIAL: NCT05298098
Title: Impact of Hypertonic Saline Solution on Acute Decompensated Heart Failure
Acronym: HSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSS-ADHF
Record Dates: First submitted 2022-01-17; First posted 2022-03-28 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Hypertonic Saline Solution; Renal Dysfunction; Diuretic
MeSH Terms: conditions — Renal Insufficiency | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Intervention Model Description: The present study is a single-center, randomized, double-blind, placebo-controlled trial performed in a tertiary hospital. It designed to evaluate the effects of the administration of hypertonic saline solution (NaCl 10%) + furosemide to patients with decompensated heart failure.
  Population:
  This study will include adult patients admitted in the emergency department for ADHF
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertonic Saline Solution (Active Comparator): 50 ml of intravenous Hypertonic Saline Solution over 1 hour + 250mg of IV furosemide over 1 hour
  Interventions: Drug: Hypertonic Saline Solution
- 5% Dextrose solution (Placebo Comparator): 50ml of 5% Dextrose solution over 1 hour + 250mg of IV furosemide over 1 hour
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hypertonic Saline Solution — Patients receive intravenous infusion of HSS (50ml of 10% NaCl) + Furosemide ( 250mg of furosemide) administered over one hour twice a day.
  Other Names: Hypertonic Saline
  Arms: Hypertonic Saline Solution
Drug: Placebo — Patients receive intravenous infusion of 5% Dextrose Solution (50ml of Dextrose 5%) + Furosemide (250mg of furosemide) administered over one hour twice a day.
  Arms: 5% Dextrose solution

SUMMARY:
Acute decompensated heart failure (HF) is one of the most common cardiologic issues in emergency departments.

Loop diuretics have long been recognized as the key for the treatment of Acute Decompensated Heart Failure (ADHF).However, chronic treatment with diuretics may limit their response and deteriorates the renal function. The hypertonic saline solution (HSS) has been proposed in recent years as an adjunctive therapy for intravenous loop diuretics to improve or restore their initial pharmacological efficacy.

In this study the investigators will evaluate the effectiveness of HSS as an adjunct to i.v. furosemide in patients admitted for AHF with renal dysfunction

DETAILED DESCRIPTION:
In the era of the emergence of novel therapies for advanced Chronic Heart Failure , the use of HSS as a therapeutic adjunct to i.v. loop diuretics still needs to be explored on a larger scale, in particular in patients with renal dysfunction.

The objective of this study is: to evaluate the effectiveness of HSS as an adjunct to i.v. furose¬mide in patients admitted for AHF with renal dysfunction.

* Patients receive intravenous infusion of HSS (50ml of 10% NaCl) + Furosemide ( 250mg of furosemide) administered over one hour twice a day.
* Patients receive intravenous infusion of 5% Dextrose Solution (50ml of Dextrose 5%) + Furosemide (250mg of furosemide) administered over one hour twice a day.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 18 years of age or older
* ADHF with congestive symptoms, laboratory(BNP) and echocardiographic criteria
* NYHA ≥II(New York Heart Association functional classification)
* Creatinine clearance≤60ml/mn (MDRD) or level of creatinine >150 µg/ml)
* BNP levels on admission ≥400 pg/mL

Exclusion Criteria:

* age < 18 years
* NYHA class < II
* Patients with acute coronary syndrome, pulmonary thromboembolism, cardiac tamponade, pericarditis, those on dialysis; patients with chronic liver disease, pleuropneumonia, cerebral vascular disease, cancer, uncompensated diabetes, patients requiring pacemaker and concomitant other important comorbidity
* Signs of hemodynamic instability, respiratory distress, coma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Length of Hospital Stay | 1 week
  The period during which the patient is hospitalized
In-hospital mortality | 1 week
  Death occuring during hospitalization
Renal Function Impairement | 1 week
  Deterioration of renal function during hospital stay
Need for inotropic drugs | 1 week
  Hemodynamic instability requiring the introduction of inotropic drugs

SECONDARY OUTCOMES:
30 day Mortality | 30 days
  Death occurring during the 30 days following discharge
Need for Renal Replacement Therapy | 1 week
  Severe Impairment of renal function requiring urgent hemodialysis
Hospital Readmission | 30 days
  Hospital readmission for acute heart failure during the 30 days following discharge

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, Professor, Principal Investigator — University of Monastir
Locations (1):
- Emergency department of university hospital Fattouma Bourguiba of Monastir Monastir, Monastir Tunisia, Monastir, Tunisia